CLINICAL TRIAL: NCT00099736
Title: Efficacy and Safety of FTY720 in Patients Who Receive a Kidney Transplant
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CFTY720A0125; CFTY720 0125 (Other: Sponsor); CFTY7200125 (Other: Sponsor)
Record Dates: First submitted 2004-12-17; First posted 2004-12-20 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Kidney Transplantation
Keywords: Kidney, transplantation, rejection, immunosuppression
MeSH Terms: conditions — Rejection, Psychology | interventions — Fingolimod Hydrochloride; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- FTY720 5 mg + reduced-dose Neoral (RDN) + corticosteroids, (Experimental)
  Interventions: Drug: FTY720 5 mg + reduced-dose Neoral (RDN) + corticosteroids
- FTY720 2.5 mg + full dose Neoral (FDN) + corticosteroids (Experimental)
  Interventions: Drug: FTY720 2.5 mg + full dose Neoral (FDN) + corticosteroids
- MMF 2 g + full-dose Neoral (FDN) + corticosteroids (Experimental)
  Interventions: Drug: MMF 2 g + full-dose Neoral (FDN) + corticosteroids

INTERVENTIONS:
Drug: FTY720 5 mg + reduced-dose Neoral (RDN) + corticosteroids — FTY720 5 mg + reduced-dose Neoral (RDN) + corticosteroids
  Arms: FTY720 5 mg + reduced-dose Neoral (RDN) + corticosteroids,
Drug: FTY720 2.5 mg + full dose Neoral (FDN) + corticosteroids — FTY720 2.5 mg + full dose Neoral (FDN) + corticosteroids
  Arms: FTY720 2.5 mg + full dose Neoral (FDN) + corticosteroids
Drug: MMF 2 g + full-dose Neoral (FDN) + corticosteroids — mycophenolate mofetil (MMF) + full-dose Neoral (FDN) + corticosteroids
  Arms: MMF 2 g + full-dose Neoral (FDN) + corticosteroids

SUMMARY:
The efficacy and safety of FTY720 is being evaluated in patients who receive a kidney transplant.

ELIGIBILITY:
Inclusion Criteria:

* First kidney transplantation
* Male and female patients
* Between 18 and 65 years old

Exclusion Criteria:

* Patients in need of multiple organ transplants

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 696 (Actual)
Dates: Start 2003-05-07; Primary Completion 2005-09-19 (Actual); Study Completion 2005-09-19 (Actual)

PRIMARY OUTCOMES:
IA, IB, IIA, IIB, III, or humoral rejection diagnosed by biopsy according to Banff 97 criteria within 12 months post transplant
permanent resumption of dialysis within 12 months post transplant
surgical removal of graft within 12 months post transplant
death within 12 months post transplant
withdrawal of consent, death, or lost to follow up within 12 months post transplant

SECONDARY OUTCOMES:
FEV1 , FVC, FEV1/FVC, DLCO and FEF 25%-75% at day 28, months 6 and 12
serum creatinine
cystatin C at months 3, 6, and 12
proteinuria at day 28, months 6 and 12
absolute lymphocyte count at screening, baseline, day 1, 7, 14, and 28, months 2, 3, 6, 9, and 12

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (39):
- United States (39):
  - Phoenix, Arizona
  - Los Angeles, California
  - Palo Alto, California
  - San Francisco, California
  - Denver, Colorado
  - New Haven, Connecticut
  - Tampa, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Des Moines, Iowa
  - Portland, Maine
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Minneapolis, Minnesota
  - Rochester, Minnesota
  - Omaha, Nebraska
  - Livingston, New Jersey
  - Hawthorne, New York
  - Chapel Hill, North Carolina
  - Durham, North Carolina
  - Cleveland, Ohio
  - Toledo, Ohio
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Dallas, Texas
  - Galveston, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Fairfax, Virginia
  - Richmond, Virginia
  - Madison, Wisconsin
  - Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Tedesco-Silva H, Pescovitz MD, Cibrik D, Rees MA, Mulgaonkar S, Kahan BD, Gugliuzza KK, Rajagopalan PR, Esmeraldo Rde M, Lord H, Salvadori M, Slade JM; FTY720 Study Group. Randomized controlled trial of FTY720 versus MMF in de novo renal transplantation. Transplantation. 2006 Dec 27;82(12):1689-97. doi: 10.1097/01.tp.0000251718.95622.b3. PMID 17198261